CLINICAL TRIAL: NCT02792023
Title: Usefulness of Fecal Immunochemical Test in the Diagnosis Algorithm of Iron Deficiency Anemia.
Brief Title: Usefulness of Fecal Immunochemical Test in Iron Deficiency Anemia (IDAFIT)
Acronym: IDAFIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario de Canarias (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FIT-Iron deficiency anemia
Record Dates: First submitted 2016-05-20; First posted 2016-06-07 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Immunochemical occult blood test
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy; Gastroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Colonoscopy followed by upper endoscopy (Other): In case of a positive immunochemical fecal occult blood test result, colonoscopy will be the first examination
  Interventions: Other: Immunochemical fecal occult blood test; Device: Colonoscopy; Device: Upper endoscopy
- Upper endoscopy followed by colonoscopy (Other): In case of a negative immunochemical fecal occult blood test result, upper endoscopy will be the first examination
  Interventions: Other: Immunochemical fecal occult blood test; Device: Colonoscopy; Device: Upper endoscopy

INTERVENTIONS:
Other: Immunochemical fecal occult blood test — Participants will be provided with a single immunochemical fecal occult blood test. Participants will introduce a small sample of feces inside and bring the test to the hospital
Device: Colonoscopy — A colonoscopy (procedure performed using a scope design to examine the large bowel) will be offered to the participants
Device: Upper endoscopy — An upper endoscopy (procedure performed using a scope to examine the upper digestive tract) will be offered to the participants

SUMMARY:
Prospective study to test whether the immunochemical fecal occult blood test (FIT) for colorectal cancer (CRC) helps to prioritize patients with iron deficiency anemia for colonoscopy.

DETAILED DESCRIPTION:
This is a multicenter (two centers), prospective study to test the accuracy of FIT for CRC detection in patients with severe IDA and its potential value for prioritizing colonoscopy.

An appointment with a gastroenterologist will be scheduled for patients with IDA referred for upper gastrointestinal endoscopy or colonoscopy. The gastroenterologist will check the inclusion and exclusion criteria. Eligible patients will sign the informed consent to carry out the following procedures:

1. Blood analysis to rule out celiac disease (anti-transglutaminase IgA antibodies and IgA).
2. A quantitative fecal immunological test (FIT: OC-Sensor ®) will be provided.
3. An appointment for colonoscopy and gastroscopy will be provided after completion of the FIT in all patients. During gastroscopy, duodenal biopsies from the second portion of the duodenum and duodenal bulb will be taken to rule out celiac disease. Biopsies from the stomach will be also taken to assess helicobacter pylori infection.
4. In patients with severe anemia colonoscopy and upper endoscopy will be prioritized (<20 days) (primary outcome).
5. Patients with colonoscopy and gastroscopy without significant lesions, will be scheduled for the performance of a capsule endoscopy.
6. Endoscopists will be blind for the FIT results.
7. the following information will be collected: consumption of acetylsalicylic acid, non steroidal anti inflammatory drugs, oral anticoagulants, corticosteroids and proton pump inhibitors (PPI). In the case of patients receiving treatment with PPIs, they will be removed 15 days before the completion of the FIT and not resumed until the performance of the upper endoscopy.

The hypothesis of the study is that one-time FIT is a useful tool for increasing the efficiency of colonoscopy and can be used to prioritize outpatient colonoscopy in patients with IDA. In order to calculate the sample size required for the study, the investigators have assumed that FIT is positive in 25% of cases with iron deficiency anemia and 20% of them would have an advanced colorectal neoplasia at colonoscopy whereas only 10% of advanced colorectal neoplasias would be found in the remaining 75% patients with a negative FIT. Considering a type I error (alpha) of 5%, a power of 80% and a percentage of losses of 15%, 550 patients will be necessary to include. The investigators estimate that approximately 15% of these patients (n=83) will have severe anemia.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive outpatients with iron deficiency anemia (Hemoglobin < 13 g/dl in males and 12 g/dl in females) referred for upper endoscopy and/or colonoscopy.
* To sign the informed consent.

Exclusion Criteria:

* < 18 years
* Pregnancy
* Personal history of inflammatory bowel disease
* Gastric / duodenal ulcer or gastrointestinal neoplasia
* Family history of hereditary CRC (Lynch Syndrome or familial adenomatous polyposis)
* Rectal bleeding / hematochezia
* Gastroscopy / colonoscopy / endoscopy capsule in the previous 5 years
* Patients not candidates for endoscopic studies because a low performance status
* Previous abdominal surgery
* Refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2016-06-30 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
The number of patients with colorectal cancer among those with a positive immunochemical fecal test (Positive predictive value) | one year
  In order to calculate the positive predictive value, the number of patients with events (colorectal cancers) will be divided among the number of positive immunochemical fecal tests

SECONDARY OUTCOMES:
The number of patients with a significant lesion among those with a positive immunochemical fecal test (Positive predictive value) after the colonoscopy and after the upper endoscopy | one year
  In order to calculate the positive predictive value, the number of patients with a significant lesion (i.e. colorectal cancer, advanced adenoma, inflammatory bowel disease, angiodysplasia, gastric cancer, watermelon stomach, gastric/duodenal ulcer, ampulloma, erosive gastritis/duodenitis) will be divided among the number of positive immunochemical fecal tests.
The number of patients without a significant lesion among those with a negative immunochemical fecal test (negative predictive value) after the colonoscopy and after the upper endoscopy | one year
  In order to calculate the negative predictive value, the number of patients without a significant lesion will be divided among patients with a negative immunochemical fecal test

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Quintero, MD, PhD, Study Director — Hospital Universitario de Canarias
Locations (1):
- Digestive Service, Huc, San Cristóbal de La Laguna, S/C de Tenerife, Spain

REFERENCES:
- [Background] James MW, Chen CM, Goddard WP, Scott BB, Goddard AF. Risk factors for gastrointestinal malignancy in patients with iron-deficiency anaemia. Eur J Gastroenterol Hepatol. 2005 Nov;17(11):1197-203. doi: 10.1097/00042737-200511000-00008. PMID 16215432
- [Background] Hamilton W, Lancashire R, Sharp D, Peters TJ, Cheng KK, Marshall T. The importance of anaemia in diagnosing colorectal cancer: a case-control study using electronic primary care records. Br J Cancer. 2008 Jan 29;98(2):323-7. doi: 10.1038/sj.bjc.6604165. Epub 2008 Jan 22. PMID 18219289
- [Background] Quintero E, Castells A, Bujanda L, Cubiella J, Salas D, Lanas A, Andreu M, Carballo F, Morillas JD, Hernandez C, Jover R, Montalvo I, Arenas J, Laredo E, Hernandez V, Iglesias F, Cid E, Zubizarreta R, Sala T, Ponce M, Andres M, Teruel G, Peris A, Roncales MP, Polo-Tomas M, Bessa X, Ferrer-Armengou O, Grau J, Serradesanferm A, Ono A, Cruzado J, Perez-Riquelme F, Alonso-Abreu I, de la Vega-Prieto M, Reyes-Melian JM, Cacho G, Diaz-Tasende J, Herreros-de-Tejada A, Poves C, Santander C, Gonzalez-Navarro A; COLONPREV Study Investigators. Colonoscopy versus fecal immunochemical testing in colorectal-cancer screening. N Engl J Med. 2012 Feb 23;366(8):697-706. doi: 10.1056/NEJMoa1108895. PMID 22356323
- [Background] Quintero E, Carrillo M, Gimeno-Garcia AZ, Hernandez-Guerra M, Nicolas-Perez D, Alonso-Abreu I, Diez-Fuentes ML, Abraira V. Equivalency of fecal immunochemical tests and colonoscopy in familial colorectal cancer screening. Gastroenterology. 2014 Nov;147(5):1021-30.e1; quiz e16-7. doi: 10.1053/j.gastro.2014.08.004. Epub 2014 Aug 13. PMID 25127679
- [Background] Rodriguez-Alonso L, Rodriguez-Moranta F, Ruiz-Cerulla A, Lobaton T, Arajol C, Binefa G, Moreno V, Guardiola J. An urgent referral strategy for symptomatic patients with suspected colorectal cancer based on a quantitative immunochemical faecal occult blood test. Dig Liver Dis. 2015 Sep;47(9):797-804. doi: 10.1016/j.dld.2015.05.004. Epub 2015 May 15. PMID 26055489
- [Background] Cubiella J, Salve M, Diaz-Ondina M, Vega P, Alves MT, Iglesias F, Sanchez E, Macia P, Blanco I, Bujanda L, Fernandez-Seara J. Diagnostic accuracy of the faecal immunochemical test for colorectal cancer in symptomatic patients: comparison with NICE and SIGN referral criteria. Colorectal Dis. 2014 Aug;16(8):O273-82. doi: 10.1111/codi.12569. PMID 24456168